CLINICAL TRIAL: NCT01568918
Title: The Use of an Uroselective Alpha-1-antagonist to Reduce the Incidence and Duration of Postoperative Urinary Retention Following Spine Surgery
Brief Title: Use of Tamsulosin to Reduce the Incidence and Duration of Postoperative Urinary Retention Following Spine Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow recruitment and enrollment
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michelle J. Clarke, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 11-006704
Record Dates: First submitted 2012-03-13; First posted 2012-04-02 (Estimated); Results first posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Postoperative Urinary Retention
MeSH Terms: interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tamsulosin (Experimental): Participants randomized to this arm will receive 0.4 mg/day tamsulosin hydrochloride from 5 days prior to the operation until hospital discharge.
  Interventions: Drug: Tamsulosin hydrochloride
- Placebo (Placebo Comparator): Participants randomized to this arm will receive a daily placebo capsule matching the active study drug from 5 days prior to the operation until hospital discharge.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tamsulosin hydrochloride — Participants will receive 0.4 mg/day tamsulosin hydrochloride from 5 days prior to the operation until hospital discharge.
  Other Names: Flomax; Flomaxtra; Contiflo XL; Urimax
  Arms: Tamsulosin
Other: Placebo — The placebo capsule matching the active study drug will be given daily from 5 days prior to the operation until hospital discharge.
  Arms: Placebo

SUMMARY:
Postoperative urinary retention is a frequent complication of spinal surgeries and impacts a large portion of this population which results in increased morbidity as a result of increased number of catheterizations, urinary tract infections (UTIs) and prolonged hospital stays. With the addition of Tamsulosin, the investigators would anticipate a reduction in the incidence and duration of postoperative urinary retention and therefore a reduction in morbidity related to treatment of urinary retention as well as shortened hospital stays.

DETAILED DESCRIPTION:
Decompressive laminectomy and spinal fusion procedures are among the most common neurosurgical procedures performed. Postoperative urinary retention (POUR) is a frequent complication of such surgeries and impacts a large proportion of this population resulting in multiple intermittent bladder catheterizations for bladder decompression, increased incidence of bacteremia, increased incidence of UTIs, and prolonged hospital stays. Use of a uroselective alpha-1-adrenergic receptor antagonist, such as tamsulosin, in the perioperative period (medication started five days prior to surgery and taken until hospital discharge) could reduce both the incidence and duration of postoperative urinary retention, resulting in shorter hospital stays and decreased healthcare costs.

ELIGIBILITY:
Inclusion Criteria

* ≥ 35 years (Males & Females)
* Cervical Laminectomy
* Cervical Posterior Fusion
* Cervical Anterior/Posterior Fusion
* Lumbar Laminectomy
* Lumbar Posterolateral Fusion
* Lumbar Interbody Fusion

Exclusion Criteria

* < 35 years
* Cervical Anterior Discectomy and Fusion
* Cervical Anterior Corpectomy
* Cervical Posterior Discectomy
* Cervical Foraminotomy
* Lumbar Discectomy (METRx or Open)
* Lumbar Foraminotomy
* Lumbar Anterior Fusion
* Myelopathy with bladder dysfunction
* Patients currently taking an alpha-antagonist
* Patients with history of allergy or sensitivity to tamsulosin or other alpha-antagonist (alfuzosin, doxazosin, prazosin, terazosin, tamsulosin, and phenoxybenzamine)
* History of prostatectomy or urologic surgery involving the bladder or urethra
* Severe liver disease or end-stage renal disease
* Patients taking strong inhibitors of CYP3A4 (ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir/ritonavir, lopinavir/ritonavir, and conivaptan)
* Patients with a mental disability
* Prisoners

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Clarke, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials website — https://clinicaltrials.gov

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tamsulosin | Placebo
Started | 39 | 51
Completed | 39 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tamsulosin | Placebo | Total
Number analyzed (Participants) | 39 | 51 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.04 (10.36) | 63.59 (9.91) | 62.47 (10.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 20 | 35
  Male | 24 | 31 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 39 | 51 | 90
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 39 | 51 | 90
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 39 | 51 | 90

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Postoperative Urinary Retention
Description: Post operative urinary retention (POUR) will be defined as any of the following:
  1) Estimated post-void residual (PVR) volume of urine greater than or equal to 300 mL; 2) Estimated retention urine volume of greater than or equal to 500 mL in patients unable to void; 3) Patients experiencing discomfort or distension and unable to void with lesser residual urine volume than 500 ml.
Time Frame: participants will be followed for the duration of the hospital stay, an expected average of 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 39 | 51
Participants | 11 | 20

2. Secondary Outcome: Duration of Postoperative Urinary Retention
Description: The neurosurgical team will decide if an indwelling urinary catheter will be used. Time of indwelling catheter removal after surgery will serve as time zero for beginning calculation of postoperative urinary retention duration if the patient later requires in and out straight catheterization. For patients without an indwelling catheter, the time patients leave the operating room will serve as time zero. Urinary retention will be considered resolved after two consecutive post-void residual urine scans have demonstrated less than 300 ml residual urine volume in a patient spontaneously voiding.
Time Frame: participants will be followed for the duration of the hospital stay, an expected average of 5 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 39 | 51
days | 3.42 (0.932) | 3.52 (1.210)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to first follow-up postop (approximately 3 months) on all participants.
Arm/Group | Tamsulosin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/51
Other Adverse Events (participants affected / at risk) | 0/39 | 1/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tamsulosin (N=39) | Placebo (N=51)
Lower Extremity Edema (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Terminated study due to slow recruitment and enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-02-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT01568918/Prot_SAP_000.pdf